CLINICAL TRIAL: NCT01727232
Title: Efficacy and Safety of Rituximab Given at Fixed Dose (1000 mg on Days 1 and 15) Compared to the Standard Regimen in Adult's Immune Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Dr Mahévas Matthieu, MD, MD, Henri Mondor University Hospital
Other Study IDs: Mondor-Rituxcompare
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; Rituximab; Efficacy; Anti-CD20; Regimen
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard regimen: Patients received the standard regimen (i.e 4 weekly infusions of 375 mg/m2)of rituximab
- Rheumatoid arthritis regimen: Patients received the RA regimen (i.e two infusions of 1000 mg, 2 weeks apart) of rituximab

SUMMARY:
The aim of this large French multicentric retrospective study was to compare the efficacy and safety of two (the standard and the Rheumatoid arthritis) rituximab regimens in adult's immune thrombocytopenia .

DETAILED DESCRIPTION:
Every adult (age ≥ 18 years) seen in one of the 3 participating centre (dijon, Marseille, Mondor) over a 7-year period (2005-2012) with a definite diagnosis of primary ITP according to the American Society Hematology guidelines who received RTX regardless the regimen could be included.

ELIGIBILITY:
Inclusion Criteria:

* Primary ITP
* Age > 18 years

Exclusion Criteria:

* Secondary ITP
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary ITP patients treated with standard or RA regimen were retrospectively included in the observationnal study.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study was to assess the response rate to treatment 1 year after the first rituximab infusion. | one year
  A complete response (CR) was defined as a platelet count >100 x 109/l and a response (R): by a platelet count >30 x 109/l with a least a doubling of the baseline value without any rescue intervention within 8 weeks before assessment, and no response (NR) was defined as a platelet count lower than 30 x 109/

SECONDARY OUTCOMES:
The response rate 3months, and at the last follow-up after the first rituximab infusion. Variable associated with RTX response. | 3 months, one year, last follow-up